CLINICAL TRIAL: NCT03533868
Title: Reaching 90% Target of HIV Viral Suppression: The Role of Point-of-Care Viral Load Monitoring in Resource-Constrained Settings in Nigeria
Brief Title: Reaching 90% HIV Suppression: The Role of POC Viral Load Monitoring in Nigeria
Acronym: POC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Jos University Teaching Hospital (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Phyllis Kanki, Professor of Immunology & Infectious Diseases, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CDC-CGH-2018-059
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: HIV/AIDS
Keywords: Point-of-care; Viral load monitoring; Nigeria
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to have their viral load monitored by either the standard of care or point-of-care method at their follow-up clinical visits up to 12 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (SOC) (No Intervention): Patients in this arm will have their viral load monitored using the standard of care method, using the Roche Cobas TaqMan HIV-1® v2 (Roche) assay.
- Point-of-care (POC) (Experimental): Patients in this arm will have their follow-up viral loads (after baseline) monitored using a Point-of-care viral load monitoring test, the Cepheid Xpert HIV-1 Viral Load assay.
  Interventions: Diagnostic Test: Point-of-care viral load monitoring test

INTERVENTIONS:
Diagnostic Test: Point-of-care viral load monitoring test — For enumerating viral load for patients in the POC arm, we will use the Cepheid Xpert® HIV-1 Viral Load test, a quantitative assay with a quantification range of 40 to 10,000,000 copies/mL. Based on the GeneXpert® technology, Xpert HIV-1 VL automates the test process, including RNA extraction, purification, reverse transcription and cDNA real-time quantitation in one fully integrated cartridge. The pre-loaded disposable single-use cartridges provide a visual read-out within 90 minutes. The assay requires 1 mL of plasma using a precision pipette (1.2 mL using a transfer pipette).
  Arms: Point-of-care (POC)

SUMMARY:
The UNAIDS 90-90-90 goals represents an ambitious strategy to end the acquired immunodeficiency syndrome (AIDS) epidemic by 2020 [UNAIDS, 2015]. While viral load (VL) quantification is the gold standard of HIV treatment monitoring, it is only routinely available and employed in resource-rich countries. The use of an affordable, reliable, point-of-care (POC) VL assay has been considered a "game-changer", where increased access, minimal lab worker training, and same day results could be addressed in a single solution. To date, POC VL assays have been evaluated by their manufacturers with reference panels of samples with some in-country laboratory evaluations. While these are appropriate and critical first steps, it is also important to evaluate the impact of this new technology against the standard of care (SOC) method of VL monitoring in an actual resource-limited setting.

Nigeria has the second highest burden of HIV in the world, with an estimated 3.2 million infected and serves as a relevant setting for testing feasibility and efficacy of POC VL monitoring [UNAIDS, 2016]. In order to present the case for implementing the use of POC VL testing across Nigeria, data on the acceptability, feasibility and efficacy of using POC testing for VL monitoring are needed. To address this need, the investigators have designed a randomized controlled trial comparing POC VL to monitoring to the SOC, which follows the Nigerian National Guidelines, to provide operational evidence for implementation of POC VL testing in Nigeria. This trial is aimed at testing the hypothesis that using POC versus SOC VL monitoring in HIV-infected patients newly initiating ART will improve overall ART outcomes, increase ART adherence and program retention rates, and result in faster switches to second-line treatment of patients failing first-line ART.

DETAILED DESCRIPTION:
The investigators will conduct an un-blinded randomized implementation trial comparing POC VL monitoring, using the Cepheid Gene Xpert HIV-1 VL®, to SOC VL monitoring, using the Roche AmpliPrep/COBAS Taqman system. The trial will be conducted at two sites in Plateau State, Nigeria.

ART-naïve patients initiating ART will be randomized on a 1:1 basis to the SOC VL monitoring control arm or the POC VL monitoring arm. VL monitoring will occur according to the current Nigerian ART guidelines-recommended algorithm, with the addition of a baseline VL test. For the month 6 and 12 visits, patients that are enrolled in the POC VL monitoring arm will be provided their VL results. Participants in the SOC arm will receive their Roche VL test results after the results become available per SOC protocol. All other aspects of their HIV care and treatment will be identical to services that they would normally receive at these treatment centers.

The investigators will follow all patients up through their Month 12 follow-up visit. At trial exit, the investigators will ask patients, caregivers of patients under the age of 18 years, and providers for their participation in surveys on the operational performance and acceptability of the POC versus SOC VL monitoring. Following that time point, the patients will continue receiving HIV care and treatment utilizing the SOC procedures for the clinic.

ELIGIBILITY:
Inclusion Criteria:

-All HIV-infected patients newly initiating ART

Exclusion Criteria:

* Previous ARV experience
* Pregnant

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with VL<1000 copies/mL at month 12 post-initiation of ART (range 11-15 months) in SOC VL versus POC VL | 12 months (range 11-15 months)
  Proportion of patients that have undetectable viral load at the end of observation (month 12) will be compared by treatment arm

SECONDARY OUTCOMES:
Difference in ART adherence patterns in patients in the SOC versus POC VL arms | From ART initiation to month 12
  Average percent adherence will be computed using patient refill data that are stored electronically. The average will be calculated as number of days supplied over total days in the given time interval, adjusting for amount of medication that should remain since last refill, computed based on amount supplied during the previous visit minus the number of days since the last visit.
Difference in loss to follow-up rates by 12 months post-initiation of ART between patients monitored with SOC versus POC VL arms | Month 12
  LTFU at month 12 is defined as not having made any refill pick-ups or clinical visits since 9-month post-initiation of ART.
Impact of trial site on differences in virologic suppression rates within patients receiving SOC VL monitoring | Month 12
  Comparison of data from two different trial sites
Difference in time from ART initiation to the confirmation of virologic failure in SOC versus POC VL monitoring arms | ART Initiation to Month 12
  Subset analysis in those that experienced virologic failure (confirmed)
Difference in time from ART initiation to switch to 2L treatment in patients in VF in SOC versus POC VL monitoring arms | ART Initiation to Month 12
  Subset analysis in those that experienced virologic failure (confirmed)
Difference in time from specimen collection to availability of VL results in patient charts in SOC versus POC VL monitoring arms | All follow-up visits at which VL monitored up to Month 12
  Comparison of time from specimen collection to the time the result is entered into the patient chart by treatment arm
Difference in time from specimen collection to delivery of VL results to patient in SOC versus POC VL monitoring arms | All follow-up visits at which VL monitored up to Month 12
  Comparison of time from specimen collection to the time the result is verbally conveyed to the patient by their clinician by treatment arm
Difference in time from lab confirmation of first unsuppressed VL to adherence counseling provided and switch to 2L in SOC versus POC VL monitoring arms | All follow-up visits at which VL monitored up to Month 12
  Subset analysis in those that experienced virologic failure (confirmed)
Difference in HIV DRM patterns in patients failing 1L ART in the SOC versus POC VL monitoring arm | Month 12
  Subset analysis in those that experienced virologic failure (confirmed)
Health care worker (HCW) satisfaction level with POC versus SOC VL monitoring | Month 12
  Health care workers will complete a standardized survey querying about their satisfaction with the POC assay. The survey uses a scale measuring agreement level. The scale ranges from 0 to 5 where 0=not applicable, 1=strongly disagree and 5=strongly agree
POC VL arm patient satisfaction with POC vs SOC VL testing | Month 12
  POC VL arm patients will be queried using a standardized survey about their satisfaction with the POC VL assay. The survey uses a scale measuring agreement level. The scale ranges from 0 to 5 where 0=not applicable, 1=strongly disagree and 5=strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Phyllis Kanki, DVM, DSc, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (2):
- Nigeria (2):
  - Jos University Teaching Hospital, Jos, Plateau State
  - Comprehensive Health Care Centre, Zamko, Zamko, Plateau State

IPD SHARING:
Plan to Share IPD: Yes
The study data set from the proposed trial, stripped of all identifying information and anonymized to protect patient confidentiality, will be available upon request within 30 months of the end of data collection.
Supporting Information: Study Protocol, SAP
Time Frame: Within 30 months of the end of data collection
Access Criteria: Reasonable request via secondary data use application per review of project Principal Investigators.

REFERENCES:
- [Background] Fonjungo PN, Boeras DI, Zeh C, Alexander H, Parekh BS, Nkengasong JN. Access and Quality of HIV-Related Point-of-Care Diagnostic Testing in Global Health Programs. Clin Infect Dis. 2016 Feb 1;62(3):369-374. doi: 10.1093/cid/civ866. Epub 2015 Sep 30. PMID 26423384
- [Background] Fonjungo PN, Osmanov S, Kuritsky J, Ndihokubwayo JB, Bachanas P, Peeling RW, Timperi R, Fine G, Stevens W, Habiyambere V, Nkengasong JN. Ensuring quality: a key consideration in scaling-up HIV-related point-of-care testing programs. AIDS. 2016 May 15;30(8):1317-23. doi: 10.1097/QAD.0000000000001031. PMID 26807969
- [Derived] Chaplin B, Agbaji O, Reyes Nieva H, Olatunde B, Chang C, Mitruka K, Sule H, Dajel T, Zee A, Ahmed ML, Ahmed I, Okonkwo P, Rawizza H, Kanki P. Timeliness of Point-of-Care Viral Load Results Improves Human Immunodeficiency Virus Monitoring in Nigeria. Clin Infect Dis. 2023 Feb 8;76(3):e671-e680. doi: 10.1093/cid/ciac609. PMID 35872644
- [Derived] Chang C, Agbaji O, Mitruka K, Olatunde B, Sule H, Dajel T, Zee A, Ahmed ML, Ahmed I, Okonkwo P, Chaplin B, Kanki P. Clinical Outcomes in a Randomized Controlled Trial Comparing Point-of-Care With Standard Human Immunodeficiency Virus (HIV) Viral Load Monitoring in Nigeria. Clin Infect Dis. 2023 Feb 8;76(3):e681-e691. doi: 10.1093/cid/ciac605. PMID 35867672
- [Derived] Meloni ST, Agbaji O, Chang CA, Agaba P, Imade G, Oguche S, Mukhtar A, Mitruka K, Cox MH, Zee A, Kanki P. The role of point-of-care viral load monitoring in achieving the target of 90% suppression in HIV-infected patients in Nigeria: study protocol for a randomized controlled trial. BMC Infect Dis. 2019 May 2;19(1):368. doi: 10.1186/s12879-019-3983-6. PMID 31046695
- See also: UNAIDS. Ambitious treatment targets: writing the final chapter of the AIDS epidemic. 2015. — http://www.unaids.org/sites/default/files/media_asset/JC2670_UNAIDS_Treatment_Targets_en.pdf
- See also: WHO. The Availability and Use of HIV Diagnostics: A 2012/2013 WHO Survey in Low- and Middle-Income Countries. Geneva. 2014. — http://apps.who.int/iris/bitstream/10665/147213/1/9789241507905_eng.pdf
- See also: UNAIDS. Country factsheets: Nigeria, 2016. — http://www.unaids.org/en/regionscountries/countries/nigeria
- See also: FMOH Nigeria. National Guidelines for Prevention Treatment and Care. 2016. — http://apps.who.int/medicinedocs/documents/s23252en/s23252en.pdf

DOCUMENTS (1):
  • Informed Consent Form (2018-02-21): https://cdn.clinicaltrials.gov/large-docs/68/NCT03533868/ICF_000.pdf